CLINICAL TRIAL: NCT07178652
Title: Preeclampsia and Defective Placentation in Oocyte Donation: Importance of HLA-C and KIR
Acronym: IMMUN-OR
Status: Not yet recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Neelke De Munck, Head of the ART lab, Universitair Ziekenhuis Brussel
Other Study IDs: EC 2023-228
Record Dates: First submitted 2025-09-02; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Preeclampsia (PE) Risk; Oocyte Donation
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cheek swab for DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PE: Patients who develop PE during their pregnancy after oocyte donation.
- No PE: Patients who do not develop PE during their pregnancy after oocyte donation.

SUMMARY:
The IMMUN-OR study aims to study HLA-C/KIR combinations when looking at the risk of development of preeclampsia (PE) in pregnancies after oocyte donation. With the use of oocyte donation currently on the rise, the importance of identifying risk factors for the higher frequency of PE development is clear. Certain HLA-C/KIR combinations have already been linked to higher risk of obstetric complications. This study will look at these combinations within the specific situation of oocyte donation. This will further investigate the importance of the immunological interface when looking at PE. Participants will be chosen from a database of all the live births after oocyte donation at our center. The research team will contact the mother, child and donor. If all three agree to participate, they will be invited to our center, where the research team will take a cheek swab. This swab will then be used to isolate a DNA sample. With these samples, we can determine the HLA-C/KIR combination for each threesome. When all samples have been collected, two groups are made based off their health outcome: one group that did develop PE during their pregnancy, and one group that did not develop PE. The different HLA-C/KIR combinations will be compared, and the research team will look to discover if one combination is linked to a higher occurrence of PE development.

ELIGIBILITY:
Inclusion Criteria:

* Every live birth delivery post oocyte donation (mother, child, donor).

Exclusion Criteria:

* Unknown HLA-C/KIR typing of acceptor, donor or offspring (resumlts of all 3 parties must be present to participate.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated for oocyte donation at the Brussels IVF center.
Sampling Method: Non-Probability Sample
Enrollment: 2325 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia development. | From 20 weeks gestation until 6 weeks postpartum.
  The development of PE throughout the pregnancy conceived through oocyte donation.

SECONDARY OUTCOMES:
Development of early onset PE versus late onset PE. | From 20 weeks gestation until 6 weeks postpartum in pregnancies conceived through oocyte donation.
  The development of PE before 34 weeks gestation (= early onset PE) or after 34 weeks of gestation (= late onset PE).
Preterm PE versus Term PE or PP PE | From 20 weeks gestation until 6 weeks postpartum in pregnancies conceived through oocyte donation.
  Development of preterm PE (<37 weeks gestation), term PE (>37 weeks gestation) and postpartum PE (after birth) throughout a pregnancy conceived through oocyte donation.
Incidence of eclampsia, placental abruption, HELLP syndrome | From conception until 6 weeks postpartum in pregnancies conceived through oocyte donation.
  The occurence of eclampsia, placental abruption and HELLP syndrome in pregnancies conceived through oocyte donation.
Obstetrical complications | From conceptions until birth in pregnancies conceived through oocyte donation.
  Incidence of obstetrical complications such as gestational hypertension, IUGR, PPROM, ...
Delivery characteristics | From conception until birth in pregnancies conceived through oocyte donation.
  Details about delivery such as preterm birth, the incidence and indication for caesarean sections, neonatal birth weights, neonatal birth defects, neonatal complications, ...